CLINICAL TRIAL: NCT00399724
Title: A Multicentre, Multinational, Randomised, Open Study to Establish the Optimal Method for Initiating and Maintaining Lantus® (Insulin Glargine) Therapy Based on a Comparison of Two Treatment Algorithms to Determine Optimal Metabolic Outcomes, Safety, and Satisfaction in Subjects With Type 2 Diabetes Mellitus.
Brief Title: A Trial Comparing Lantus Algorithms to Achieve Normal Blood Glucose Targets in Subjects With Uncontrolled Blood Sugar With Type 2 Diabetes Mellitus
Acronym: AT-LANTUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_3504
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin glargine

SUMMARY:
Primary objective:

* To determine the optimal treatment algorithm for the clinical use of insulin glargine based on the incidence of severe hypoglycaemia.

Secondary objectives:

* To determine for each treatment algorithm the incidence of asymptomatic, symptomatic and nocturnal hypoglycaemia.
* To determine the difference in glycaemic control as measured by HbA1c and fasting blood glucose between the treatment algorithms.
* To determine the difference in glycaemic control as measured by HbA1c and fasting blood glucose between baseline and end of treatment.
* To obtain safety data on the use of insulin glargine in each treatment algorithm.
* To measure change in subject weight and insulin dose between baseline and end of treatment.
* To determine subject quality of life and treatment satisfaction (sub-study)

ELIGIBILITY:
Inclusion criteria:

* Subjects with Type 2 Diabetes Mellitus,
* Subjects on antidiabetic treatment (oral and/or insulin therapy) for > 6 months,
* Subjects who require a basal long-acting insulin for the control of hyperglycaemia,
* HbA1c values > 7.0% and < 12 %,
* BMI < 40 kg/m².

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7376
Dates: Start 2002-03; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Incidence of severe hypoglycaemia

SECONDARY OUTCOMES:
Incidence of any hypoglycaemia
Incidence of symptomatic hypoglycaemia
Incidence of nocturnal hypoglycaemia
Incidence of asymptomatic hypoglycaemia
Adjusted mean change in Hb1Ac (%)
Adjusted mean change in fasting blood glucose (FBG) (mg/dl)
Adjusted mean change in nocturnal blood glucose (NBG) (mg/dl)
Adjusted mean change in mean daily blood glucose (MBG) (mg/dl)
% of subjects at v12 with Hb1Ac < or = 6.5 %
% of subjects at v12 with Hb1Ac < or = 7.0 %
% of subjects at v12 with FBG < or = 100 mg/dl
Weight change (kg)
Change in insulin glargine dose v2 - v12 (IU)
Safety data
Quality of Life and treatment satisfaction before, during and at the end of treatment using the Diabetes Treatment Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Sinnassamy, MD, Study Director — Sanofi

REFERENCES:
- [Result] Davies M, Lavalle-Gonzalez F, Storms F, Gomis R; AT.LANTUS Study Group. Initiation of insulin glargine therapy in type 2 diabetes subjects suboptimally controlled on oral antidiabetic agents: results from the AT.LANTUS trial. Diabetes Obes Metab. 2008 May;10(5):387-99. doi: 10.1111/j.1463-1326.2008.00873.x. Epub 2008 Mar 18. PMID 18355327
- [Result] Davies M, Sinnassamy P, Storms F, Gomis R; AT.LANTUS Study Group. Insulin glargine-based therapy improves glycemic control in patients with type 2 diabetes sub-optimally controlled on premixed insulin therapies. Diabetes Res Clin Pract. 2008 Feb;79(2):368-75. doi: 10.1016/j.diabres.2007.09.013. Epub 2007 Nov 5. PMID 17980928
- [Result] Davies M, Storms F, Shutler S, Bianchi-Biscay M, Gomis R; ATLANTUS Study Group. Improvement of glycemic control in subjects with poorly controlled type 2 diabetes: comparison of two treatment algorithms using insulin glargine. Diabetes Care. 2005 Jun;28(6):1282-8. doi: 10.2337/diacare.28.6.1282. PMID 15920040
- [Derived] Khunti K, Srinivasan BT, Shutler S, Davies MJ. Effect of insulin glargine on glycaemic control and weight in obese and non-obese people with type 2 diabetes: data from the AT.LANTUS trial. Diabetes Obes Metab. 2010 Aug;12(8):683-8. doi: 10.1111/j.1463-1326.2010.01217.x. PMID 20590745